CLINICAL TRIAL: NCT05943106
Title: A Phase IIIb Open-Label, Single-Arm, Multi-Center, US Study of Bacillus Calmette-Guerin (BCG) Administered in Combination With Durvalumab in Adult BCG-naïve, High-risk Non-Muscle- Invasive Bladder Cancer Participants (PATAPSCO)
Brief Title: BCG in Combination With Durvalumab in Adult BCG-naïve, High-risk NMIBC Participants
Acronym: PATAPSCO
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D419JC00002
Record Dates: First submitted 2023-07-05; First posted 2023-07-13 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Non-Muscle- Invasive Bladder Cancer
Keywords: Bacillus Calmette-Guerin (BCG); BCG-naïve; immunotherapeutics; human mAb; Durvalumab; non-muscle-invasive bladder cancer (NMIBC)
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Durvalumab + BCG (Experimental): Participants will receive Durvalumab for 13 cycles every 4 weeks (q4w) for a maximum 12 months. All participants will receive BCG (supplied by the site) intravesically, as induction weekly for 6 weeks. Patients will subsequently receive BCG for maintenance for 3 weekly doses at 3,6,12,18, and up to 24 months, at the physician's discretion.
  Interventions: Biological: Durvalumab; Biological: BCG

INTERVENTIONS:
Biological: Durvalumab — Participants will receive Durvalumab via intravenous infusion from Week 1 for 13 cycles every 4 weeks (q4w) for maximum 12 months.
Biological: BCG — Participants will receive BCG via intravesical as induction weekly for 6 weeks starting at Week 1, Day 1 and subsequently for maintenance for 3 weekly doses up to 3, 6, 12, 18, and 24 months, at the physician's discretion as Standard of care.

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and efficacy profile of durvalumab + BCG (induction and maintenance) combination therapy in adult United States participants with a histologically confirmed diagnosis of high-risk non-muscle-invasive bladder cancer (NMIBC), who have received no prior systemic therapy for NMIBC, and who are BCG-naïve.

DETAILED DESCRIPTION:
This is an open-label, single-arm, multi-center, Phase IIIb US study exploring the combination of durvalumab and BCG (induction and maintenance) in participants with high-risk NMIBC.

Each participant will have screening activities up to 4 weeks before initiation of study intervention, receive study intervention for up to 24 months, followed by 3 months safety follow-up. Participants will continue to be followed up for survival until 2 years from the date of treatment initiation of the last participant enrolled in this study (approximately 42 months after first participant enrolled).

ELIGIBILITY:
Inclusion Criteria:

* BCG-naïve (defined as participants not having received prior intravesical BCG or who previously received but stopped BCG more than 3 years before study entry).
* Local histological confirmation (based on cytology and/or pathology report) of high-risk transitional cell carcinoma of the urothelium of the urinary bladder confined to the mucosa or submucosa.
* Complete resection of all Ta/T1 papillary disease prior to enrollment, with the transurethral resection of bladder tumor (TURBT) removing high-risk NMIBC (non-muscle invasive bladder cancer) performed not more than 4 months before enrollment in the study.
* No prior radiotherapy for bladder cancer.
* A life expectancy of at least 12 weeks (90 days).
* Adequate organ and marrow function
* World Health Organization/Eastern Cooperative Oncology Group performance status of 0 or 1 at screening
* No prior exposure to immune-mediated therapy of cancer
* A candidate for BCG treatment.
* Local histological confirmation (based on cytology and/or pathology report) of high-risk transitional cell carcinoma of the urothelium of the urinary bladder confined to the mucosa or submucosa. A high-risk tumor is defined as one of the following: T1 tumor; High-grade/G3 tumor; CIS.

Exclusion Criteria:

* Evidence of muscle-invasive, locally advanced, metastatic, and/or extra-vesical bladder cancer (ie, T2, T3, T4, and / or Stage IV).
* Predominantly variant histology such as micropapillary, plasmacytoid, nested, sarcomatoid, microcystic, squamous and adeno variants of UC representing > 50% of tumor tissue or other than urothelial tumors as assessed by pathology.
* Evidence of lymphovascular invasion of bladder tumor, except if treatment with BCG is deemed to be the only clinically viable treatment.
* Immediate cystectomy is indicated.
* Known or documented absolute and/or relative contraindication of adjuvant intravesical BCG treatment.
* Concurrent extravesical, non-muscle-invasive transitional cell carcinoma of the urothelium.
* History of allogenic organ transplantation. Participants with any history of allogenic stem cell transplantation are also excluded.
* Active or prior documented autoimmune or inflammatory disorders.
* Participants with hypothyroidism stable on hormone replacement.
* History of active primary immunodeficiency.
* Active infection including hepatitis B (known positive HBV/HBsAg result), HCV, or HIV 1/2 (positive HIV) antibodies.
* Current or prior use of immunosuppressive medication within 14 days before the first durvalumab dose.
* Female participants who are pregnant or breastfeeding or male or female participants of reproductive potential who are not willing to employ highly effective birth control.
* Any concurrent chemotherapy, study intervention, biologic or hormonal therapy for cancer treatment; uncontrolled intercurrent illness;
* History of another primary malignancy except for Malignancy treated with curative intent and with no known active disease ≥ 2 years; Adequately treated nonmelanoma skin cancer or lentigo maligna without evidence of disease; Adequately treated CIS without evidence of disease; Prostate cancer of stage ≤ T2cN0M0 without biochemical recurrence or progression that in the opinion of the Investigator does not require active intervention.
* Previous or concurrent treatment with potent systemic immunostimulatory agents

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-08-11 (Actual); Primary Completion 2025-06-16 (Actual); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Grade 3 or 4 Possibly related adverse events (PRAEs) | From the date of the first dose of study treatment (Day 1) until 6 months after the initiation of study treatment
  A PRAE is defined as an AE that has been assessed by the Investigator to be possibly related to study treatment. A PRAE will be included if it has onset or worsens (by Investigator report of an increase in CTCAE (common terminology criteria for adverse events) grade relative to pre-treatment) within 6 months of initiation of study intervention and it has CTCAE Grade 3 or 4 recorded within this timeframe.

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | From screening (Day -28 to -1) until 90 days following discontinuation of the last dose of study treatment (approximately 28 months)
  To further assess the safety and tolerability of durvalumab + BCG (induction and maintenance) combination therapy in high risk NMIBC participants. Number of participants with adverse events (AEs), including PRAEs, adverse events of special interest (AESIs), immune-mediated AEs, serious adverse events (SAEs), AEs resulting in treatment interruption and discontinuation will be assessed.
Percentage of patient-reported treatment tolerability symptoms assessed using specific PRO-CTCAE (Patient-Reported Outcomes- Common Terminology Criteria for Adverse Events) | Up to 24 months
  To assess patient-reported treatment tolerability in high-risk NMIBC participants treated with durvalumab + BCG (induction and maintenance) combination therapy by descriptive summary of PRO-CTCAE.
  Percentage of all dosed participants reporting each response category of each of the 19 relevant disease symptom items as measured by PRO-CTCAE. The PRO-CTCAE system, is an item bank of symptoms experienced by participants while undergoing treatment of their cancer.
Complete response rate (CRR) | At 6 months
  Complete response rate (CRR) is defined as the percentage of participants having carcinoma in situ (CIS) prior to study entry or at baseline cystoscopy who do not have CIS at 6 months.
Disease-free survival (DFS) | At 12 months and 24 months
  Disease-free survival (DFS) is defined as the time from the date of first dose of study intervention until the date of first recurrence of high-risk disease or death (by any cause in the absence of recurrence) regardless of whether the participant withdraws from therapy or receives another anticancer therapy prior to recurrence.
Overall survival (OS) | At 24 months
  Overall survival (OS) is defined as the time from the date of the first dose of study intervention to the date of death from any cause.
  The analysis will include all dosed participants. All deaths will be included regardless of whether the participant withdraws from therapy or receives another anticancer therapy.
Best overall response for health-related quality of life (HRQoL) as assessed by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 items (EORTC QLQ-C30) | Up to 24 months
  Best overall response is defined as the best response the participant achieved, based on evaluable data collected during the study period to assess disease and treatment related symptoms and HRQoL. The domains/scales of the EORTC QLQ-C30 prioritized include global HRQoL, physical functioning and fatigue. Final scores range from 0 to 100, where higher scores on the global measure of health status and functional scales indicate better health status/function, but higher scores on symptom scales represent greater symptom severity.
Best overall response for HRQoL as assessed by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Non-Muscle-Invasive Bladder Cancer 24 (EORTC QLQ-NMIBC24) | Up to 24 months
  Best overall response is defined as the best response the participant achieved, based on evaluable data collected during the study period. The domains/scales of the EORTC QLQ-NMIBC24 prioritized include urinary symptoms, intravesical treatment concerns, future perspectives and sexual functioning. Final scores range from 0 to 100, higher scores on the functioning scales (sexual functioning, sexual enjoyment) indicate better health status/function, whereas higher scores on symptom scales and individual symptom items represent greater symptom severity.

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Research Site, Phoenix, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, San Diego, California
  - Research Site, Lakewood, Colorado
  - Research Site, Hialeah, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Greenwood, Indiana
  - Research Site, Wichita, Kansas
  - Research Site, Baltimore, Maryland
  - Research Site, Hanover, Maryland
  - Research Site, Royal Oak, Michigan
  - Research Site, Troy, Michigan
  - Research Site, Syracuse, New York
  - Research Site, Cincinnati, Ohio
  - Research Site, Bala-Cynwyd, Pennsylvania
  - Research Site, Myrtle Beach, South Carolina
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home